CLINICAL TRIAL: NCT00267618
Title: Family Help Program: Primary Care Delivery by Telephone for Psychological and Behavioural Problems (Pediatric Recurrent Headache and Abdominal Pain)
Brief Title: Family Help Program: Pediatric Recurrent Headache and Abdominal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2234d; CHIR CAHR-43273
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Pediatric Recurrent Headache & Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 50% randomized to receive FHP Pain intervention
  Interventions: Behavioral: FHP Pain
- control (No Intervention): 50% randomized to receive standard/usual care for recurrent headache/abdominal pain

INTERVENTIONS:
Behavioral: FHP Pain — Evidence-based psychological and behavioural Intervention
  Arms: Treatment

SUMMARY:
The purpose of the Strongest Families (formerly Family Help Program)is to evaluate the effectiveness of the Strongest Families distance intervention compared to usual or standard care that is typically provided to children with mild to moderate Recurrent Headache/Abdominal Pain symptomology. This is a single-centre trial based at the IWK Health Centre. The primary outcome is change in diagnosis.

DETAILED DESCRIPTION:
The purpose of the Family Help Program is to deliver, primary care mental health services to children and their families in the comfort and privacy of their own home. Approximately 106 children (9-12 years of age)suffering from mild to moderate (but clinically significant) symptoms of pediatric Recurrent Headache/Abdominal Pain will be randomized.

The intervention is delivered from a distance, using educational materials (manuals, video-tapes, audio-tapes) and telephone consultation with a trained paraprofessional "coach" who is supervised by a licensed health care professional. The telephone coach delivers consistent care based on written protocols, with on-going evaluation by a professional team.

Fifty percent of the eligible participants will receive Family Help Program telephone-based treatment and 50% will be referred back to their family physician to receive standard care as determined by that physician. Those receiving standard care will be evaluated for outcome results and then compared to the Family Help treated participants. It is anticipated that Family Help treatment will be proven to be as or more effective than standard care.

ELIGIBILITY:
Inclusion Criteria:

* child 9 to 16 years of age
* child had recurrent headache and abdominal pain at least 3 times a month
* child's physical examination normal
* access to a telephone in the home
* speak and write english
* mild to moderate anxiety symptomology

Exclusion Criteria:

* child's pain due to trauma, systemic disease or disorder
* child received any psychological treatment for this or similar disorder in the past 6 months

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Diagnosis using KSADS at baseline, 120, 240 and 365 day follow-up. | baseline, 120, 240 and 365 day follow-up

SECONDARY OUTCOMES:
Symptomology frequency as evidenced by diary data; | daily during treatment; 3 weeks on follow-up at 240 & 365 day post randomization
Evaluated according to IHS criteria | baseline, 120, 240 and 365 day follow-up
Disability Measure; | weekly during treatment; baseline, 120, 240 and 365 day follow-up
Child Health Questionnaire | baseline, 120, 240 and 365 day follow-up
Economic Outcome assessment | baseline, 120, 240 and 365 day follow-up
Satisfaction measure, designed by the investigator | end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. McGrath, PhD., Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Lingely-Pottie P, McGrath PJ. A therapeutic alliance can exist without face-to-face contact. J Telemed Telecare. 2006;12(8):396-9. doi: 10.1258/135763306779378690. PMID 17227604
- [Background] McGrath PJ, Lingley-Pottie P, Emberly DJ, Thurston C, McLean C. Integrated knowledge translation in mental health: family help as an example. J Can Acad Child Adolesc Psychiatry. 2009 Feb;18(1):30-7. PMID 19270846
- [Background] Lingley-Pottie P, McGrath PJ. Telehealth: a child and family-friendly approach to mental health-care reform. J Telemed Telecare. 2008;14(5):225-6. doi: 10.1258/jtt.2008.008001. PMID 18632994
- [Background] Lingley-Pottie P, McGrath PJ. Distance therapeutic alliance: the participant's experience. ANS Adv Nurs Sci. 2007 Oct-Dec;30(4):353-66. doi: 10.1097/01.ANS.0000300184.94595.25. PMID 18025870
- [Background] Lingley-Pottie P, McGrath PJ. A paediatric therapeutic alliance occurs with distance intervention. J Telemed Telecare. 2008;14(5):236-40. doi: 10.1258/jtt.2008.080101. PMID 18632997
- See also: Family Help Program — http://www.bringinghealthhome.com/